CLINICAL TRIAL: NCT00657917
Title: Topical Treatment of Recalcitrant Ulcerative Old World Leishmaniasis With WR 279,396
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects were enrolled since the first subject completed the study 08Jun2007
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-13225
Record Dates: First submitted 2008-02-22; First posted 2008-04-14 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Cutaneous Leishmaniasis
Keywords: leishmaniasis; cutaneous; Old World; Leishmania major; Treatment
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paromomycin +Gentamicin topical cream (Experimental): WR279,396 topically twice a day for 20 days
  Interventions: Drug: Paromomycin +Gentamicin topical cream

INTERVENTIONS:
Drug: Paromomycin +Gentamicin topical cream — WR297,396 for treatment of patients with parasitologically confirmed, primarily ulcerative, Old World CL, who had either failed pentavalent antimony treatment, or who where ineligible for pentavalent antimony therapy.
  Other Names: WR279,396

SUMMARY:
The primary objective of this protocol is to treat laboratory confirmed cutaneous leishmaniasis with WR 279,396 in military health care beneficiaries. In this study "cutaneous leishmaniasis" is defined as Old World Leishmaniasis if acquired in the Southwest Central Asia/Middle East.

DETAILED DESCRIPTION:
Up to 10 volunteers, who are military health care beneficiaries, with a diagnosis of Old World cutaneous leishmaniasis who have failed pentavalent antimony or are not eligible to be treated with pentavalent antimony, will be treated with WR 279,396 (topical paromomycin-gentamicin-AQIC) twice a day for 20 days. Primary endpoint will be the appearance of complete epithelialization of each skin lesion by Day 50+/-2 weeks, or estimated 50%-99% re-epithelialization by Day 50+/-2 weeks followed by complete epithelialization by Day 100+/-2 weeks,with both categories without relapse by Day 180+/-30 days. Efficacy will be evaluated by clinical appearance assessed by study investigator and documented with photographs of the treated skin lesions. Toxicity will be evaluated by local adverse reactions and by laboratory signs of systemic toxicity.

ELIGIBILITY:
Inclusion Criteria:

Parasitologically confirmed, primarily ulcerative, Old World CL, in a patient who had either failed pentavalent antimony treatment, or who was ineligible for pentavalent antimony therapy.

* Military health care beneficiary 18 years of age or greater, unless active military in which case, 17 years is the minimum age
* Proven parasitological diagnosis by culture, PCR or microscopy in at least one skin lesion
* Lesions primarily ulcerative (i.e., not verrucous or nodular)
* Written informed consent to participate in protocol
* Negative pregnancy test within 72 hours of starting protocol
* Agrees to take precautions not to become pregnant or father a child for at least two months after completion of treatment with WR 279,396
* Cutaneous leishmaniasis acquired in Southwest Central Asia/Middle East*
* Inadequate response to treatment with pentavalent antimony or medical condition that precludes the use of pentavalent antimony

Exclusion Criteria:

* Drug intolerance: history of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides in the patient
* any leishmanial lesion on mucosal surface
* Presence of signs or symptoms of peripheral neuropathic myasthenia gravis, neuromuscular block
* Routinely taking nephrotoxic or ototoxic medications
* Disseminated disease defined as clinically significant subcutaneous nodules that are in the lymphatic drainage tract for the skin lesion with regional adenopathy > 1 cm
* Abnormal Romberg test at baseline
* Clinically significant medical problems of the kidney or liver as determined by history and by the following laboratory studies:

  * Kidney: Creatinine > 2x the upper limit of normal
  * Liver: ASTor ALT >4x the upper limit fo normal

    * This includes "L. major," "L. tropica," and "L. infantum" with over 98% of cases in U.S. military in 2002-2004 being "L. major"

      * An inadequate response to treatment with pentavalent antimony includes patients who show no or little improvement during a 15-20 day treatment course, those that initially epithelialize but later show signs of breakdown/ ulceration or develop new lesions. In general, for those with initial treatment response, would recommend waiting for approximately two months after pentavalent antimony and if lesion is not epithelialized at that time, consideration for further therapy is advised.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-12-20 (Actual); Primary Completion 2007-06-08 (Actual); Study Completion 2010-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COL Naomi Aronson, M.D., Principal Investigator — Uniformed Services Univ of the Health Sciences
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at Walter Reed Army Medical Center, Washington, DC. One subject was enrolled.
Period: Overall Study
Arm/Group | Paromomycin +Gentamicin Topical Cream
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paromomycin +Gentamicin Topical Cream
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Appearance of Complete Epithelialization of Ulcerative Lesions Caused by Old World Cutaneous Leishmaniasis With no Relapse
Description: Appearance of complete (100%) epithelialization of a skin lesion at day 50+2 weeks, or the estimated 50%-99% re-epithelialization by day 50+2 weeks followed by complete eipithelialization by day 100+2 weeks, with both categories without relapse by day 180+30 days. Ulcer measured in millimeters.
Time Frame: 180 days
Population: Ultimately, the planned statistical analysis could not be performed because only one patient was enrolled in the study.
Measure: Number; unit: Surface area in millimeters squared
Arm/Group | Paromomycin +Gentamicin Topical Cream
Number analyzed (Participants) | 1
Surface area in millimeters squared
  Screening | 2,142
  Day 20+3 | 1,488
  Day 50+14 | 1,400
  Day 180+30 (photos only) | 0

2. Secondary Outcome: Number of Relapses
Description: Evaluate the number of relapses occurring by day 180
Time Frame: 180 days
Population: Ultimately, the planned statistical analysis could not be performed because only one patient was enrolled in the study.
Measure: Number; unit: Number of relapses
Arm/Group | Paromomycin +Gentamicin Topical Cream
Number analyzed (Participants) | 1
Number of relapses | 0

3. Secondary Outcome: Safety and Tolerability (SAE's and AE's)
Description: Evaluate safety and tolerability as measured by completion of a full prescribed treatment course, treatment interruptions, SAE's and AE's
Time Frame: 180 days
Population: Ultimately, the planned statistical analysis could not be performed because only one patient was enrolled in the study.
Measure: Number; unit: Number of AE's
Arm/Group | Paromomycin +Gentamicin Topical Cream
Number analyzed (Participants) | 1
Number of AE's
  AEs Considered Related to Study Drug | 9
  AE's Not Considered Related to Study Drug | 23

ADVERSE EVENTS:
Time Frame: 180 Days
Description: Solicited and unsolicited AEs were collected throughout the 20-day treatment period. Follow-up contacts to assess efficacy and safety occurred on study days 50+14, 100+14, and 180+30.
Arm/Group | Paromomycin +Gentamicin Topical Cream
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paromomycin +Gentamicin Topical Cream (N=1)
Left calf pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to study drug
Flu-like symptoms (General disorders) | 1 (1) — Not related to study drug
Gastroenteritis (Gastrointestinal disorders) | 1 (1) — Not related to study drug
Elevated BP readings (Investigations) | 1 (1) — Not related to study drug
Right gluteal pain (General disorders) | 1 (1) — Not related to study drug
Right groin rash (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study drug
Left foot edema (Metabolism and nutrition disorders) | 1 (1) — Not related to study drug
Upper respiratory infection (Infections and infestations) | 1 (1) — Not related to study drug
Burning sensation at site (Nervous system disorders) | 1 (1) — Possibly related to study drug
Worsening pain at ulcer site (General disorders) | 1 (1) — Possibly related to study drug
Vesicle formation at ulcer site (Injury, poisoning and procedural complications) | 1 (1) — Definitely related to study drug
Intermittent tachycardia (Cardiac disorders) | 1 (1) — Not related to study drug
Blood-tinged secretions from nares (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study drug
Decreased sodium level (Investigations) | 1 (1) — Not related to study drug
Insufficient hypertension control (Vascular disorders) | 1 (1) — Not related to study drug
Cracked skin surrounding ulcer area (Skin and subcutaneous tissue disorders) | 1 (1) — Possibly related to study drug
Erosive areas around ulcer border (Skin and subcutaneous tissue disorders) | 1 (1) — Definitely related to study drug
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study drug
Rash above surrounding area of ulcer/lesion (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study drug
Blister-like formation above border of ulcer/lesion (Injury, poisoning and procedural complications) | 1 (1) — Not related to study drug
Small cut on left shin (Injury, poisoning and procedural complications) | 1 (1) — Not related to study drug
Numbness (slight) above ulcer/lesion (Nervous system disorders) | 1 (1) — Not related to study drug
Lymphadenopathy (right inguinal area) (Blood and lymphatic system disorders) | 1 (1) — Not related to study drug
Incomplete healing of ulcer/lesion (General disorders) | 1 (1) — Definitely related to study drug
Persistent lymphedema, left lower extremity (Blood and lymphatic system disorders) | 1 (1) — Not related to study drug
Dizziness (Nervous system disorders) | 1 (1) — Not related to study drug
Hyperemic left leg (Vascular disorders) | 1 (1) — Not related to study drug
Edema, left leg to mid thigh (Metabolism and nutrition disorders) | 1 (1) — Not related to study drug
Elevated percentage of monocytes in blood (Investigations) | 1 (1) — Not related to study drug
Elevated percentage of WBC in urine (Investigations) | 1 (1) — Not related to study drug
Increased drainage from wound (Surgical and medical procedures) | 1 (1) — Possibly related to study drug

LIMITATIONS AND CAVEATS:
Early termination due to only 1 patient enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No